CLINICAL TRIAL: NCT03251742
Title: Feasibility and Efficacy Of Negative Pressure Ventilation in Fontan populatioN: Cardiovascular Flow Assessment by Magnetic Resonance Imaging
Brief Title: Feasibility and Efficacy of Portable Non-invasive Negative Pressure Ventilation in Fontan Patients
Acronym: FONTAN-CMR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hayek Medical (Unknown)
Responsible Party: Principal Investigator, Pradeepkumar Charla, Clinical Fellow, University Health Network, Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Fontan0615
Record Dates: First submitted 2017-04-04; First posted 2017-08-16 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Fontan Physiology
Keywords: Fontan operation; Negative pressure ventilation; MRI

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional study designed to evaluate the immediate impact of negative pressure ventilation (NPV) in an ambulatory Fontan population using cardiovascular magnetic resonance imaging (CMR) for assessment of cardiovascular flows.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fontan patient population (Active Comparator)
  Interventions: Device: Hayek RTX ventilator
- Healthy volunteers (Sham Comparator)
  Interventions: Device: Hayek RTX ventilator

INTERVENTIONS:
Device: Hayek RTX ventilator — Negative pressure ventilation in Fontan patients.
  Other Names: Cuirass; Negative pressure ventilation

SUMMARY:
The human heart has 4 chambers: 2 collecting chambers (atria) and 2 pumping chambers (ventricles) to allow blood flow within two distinct circuits: "pulmonary" and "systemic". The pulmonary circuit directs the blood to the lungs to receive oxygen and the systemic circuit delivers oxygen-rich blood throughout the body. In children born with a single ventricle, blood from these two circuits mixes within the heart resulting in lower oxygen levels in the blood delivered to the body (cyanosis).

The Fontan procedure is a palliative surgery which bypasses the need for a ventricle to deliver blood to the lungs, as blood from the body flows passively to the lungs by a man-made connection (whereby two large body veins [cavae] are sewn to the pulmonary arteries), thereby preventing mixing of blood through restoration of two distinct circuits without mixing of blood. Although the Fontan operation effectively eliminates cyanosis and enables survival into adulthood, increased systemic venous pressure is an unavoidable systemic complication and low cardiac output (CO) is pervasive finding.

Despite excellent pediatric surgical results, the risk of late complications and death dramatically increases in the decades following Fontan surgery. A chronically low CO state secondary to decreased forward flow of blood to the lungs can result in end-organ dysfunction and shortened life expectancy. Short of heart transplantation, deemed suitable only for a minority of patients, effective therapies for low CO are largely absent. The investigators aim to investigate a novel, non-invasive, ambulatory therapy which can augment CO. Specifically, external suction is applied intermittently to the chest wall, much like a vacuum, to increase CO, called negative pressure ventilation (NPV) using a Cuirass® ventilator (Hayek Medical). Although used in patients with lung disease, the investigators' proposal is to evaluate this novel, portable, ventilation system would be the first study of its kind in adults with congenital heart disease, specifically those with a Fontan palliation.

ELIGIBILITY:
Inclusion Criteria:

* Fontan patients age > 13 years.

Exclusion Criteria:

* unable to complete MRI (pacemaker/defibrillator/retained wires, pregnancy, claustrophobia);
* evidence of Fontan failure (requiring ongoing medical / device therapy) protein-losing enteropathy, intracardiac thrombus, anatomical obstruction to the Fontan circuit;
* patent Fontan fenestration;
* oxygen saturation < 90%;
* ongoing arrhythmia;
* ejection fraction < 50% on echocardiography or CMR;
* moderate or severe valve insufficiency on echocardiography or CMR;
* Obesity (BMI >35);
* severe obstructive sleep apnea (AHI>20);
* chronic obstructive lung disease (FEV1/FVC<60%);
* severe chest wall deformities (scoliosis, kyphosis, kyphoscoliosis);
* acute or chronic kidney disease (eGFR<60)
* unable to provide informed consent.

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the NPV on cardiac output | 6-8 months
  Cardiac output will be measured in L/min/m2 using phase contrast MRI. Flow measurements will be made at baseline and with application of the device.
Efficacy of the NPV on organ perfusion | 6-8 months
  Multi organ perfusion will be measured in L/min/m2 using phase contrast MRI. Flow measurements will be made at baseline and with application of the device.

SECONDARY OUTCOMES:
Tolerability and safety of negative pressure ventilation. | 6-8 months
  Assessed by participant questionnaire rating tolerance, safety, overall satisfaction with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Wald, MD, MS, Principal Investigator — Toronto General Hospital/University Health Network; Pradeepkumar Charla, MD, MS, Study Director — Toronto General Hospital/University Health Network
Locations (1):
- Toronto General Hospital/University of Toronto., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaji S, Zafar MA, Christopher A, Saraf A, Hoskoppal A, Lanford L, Kreutzer J, Olivieri L, Alsaied T. Augmented Biphasic Breathing Using Sniff and an Oral Positive Expiratory Pressure Device (Sniff-PEP) in Fontan Patients. Pediatr Cardiol. 2025 Aug;46(6):1725-1732. doi: 10.1007/s00246-024-03598-3. Epub 2024 Jul 19. PMID 39028352